CLINICAL TRIAL: NCT05829122
Title: Sutureless Intrascleral Intraocular Lens Fixation and Modified Iris Cerclage Pupilloplasty for Aphakia and Traumatic Mydriasis
Brief Title: Sutureless Intrascleral Intraocular Lens Fixation and Modified Iris Cerclage Pupilloplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changzhou Second People's Hospital affiliated with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XinyuG
Record Dates: First submitted 2023-03-30; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-03

CONDITIONS: Aphakia; Mydriasis
Keywords: Aphakia; Mydriasis
MeSH Terms: conditions — Aphakia; Mydriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sutureless Intrascleral Intraocular Lens Fixation and Modified Iris Cerclage Pupilloplasty (Experimental)
  Interventions: Procedure: Sutureless Intrascleral Intraocular Lens Fixation and Modified Iris Cerclage Pupilloplasty

INTERVENTIONS:
Procedure: Sutureless Intrascleral Intraocular Lens Fixation and Modified Iris Cerclage Pupilloplasty — In this study, patients with various causes of pupillary dilatation were recruited, and medical records and ophthalmology examinations, including slit-lamp examination, visual acuity, corrected visual acuity, intraocular pressure, pupil diameter, pupil area, corneal endothelial cell count fundus examination, and photophobia score, were collected. Those who met the recruitment criteria underwent modified iris cerclage. The modified iris cerclage was performed by making four clear corneal incisions, suturing the iris 3-4 times consecutively between each two incisions, completing 360 degrees of iris suturing in sequence, and finally tying the knot intraocularly to complete the iris cerclage.

SUMMARY:
In this study, patients with various causes of pupillary dilatation were recruited, and medical records and ophthalmology examinations, including slit-lamp examination, visual acuity, best corrected visual acuity, intraocular pressure, pupil diameter, corneal endothelial cell count, fundus examination, and photophobia score, were collected. Those who met the recruitment criteria underwent modified iris cerclage pupilloplasty. The modified iris cerclage pupilloplasty was performed by making four clear corneal incisions, suturing the iris 3-4 times consecutively between each two incisions, completing 360 degrees of iris suturing in sequence, and finally tying the knot intraocularly to complete the iris cerclage.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of aphakia
* permanently dilated pupils
* history of phacoemulsification and pars plana vitrectomy surgeries for lens dislocation after blunt trauma

Exclusion Criteria:

* iris defects
* severe diseases such as cyclodialysis cleft, uncontrolled IOP, retinal detachment
* poorly controlled systemic diseases such as diabetes and hypertension
* corneal endothelial cell counts of <1000/mm2
* <6 months of follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
best corrected visual acuity | preoperatively
  logMAR
best corrected visual acuity | 6 months postoperatively
  logMAR
intraocular pressure | preoperatively
  mmHg
intraocular pressure | 6 months postoperatively
  mmHg
pupil diameter | preoperatively
  mm
pupil diameter | 6 months postoperatively
  mm
corneal endothelial cell count | preoperatively
  cell/mm2
corneal endothelial cell count | 6 months postoperatively
  cell/mm2

CONTACTS AND LOCATIONS:
Locations (1):
- Preoperatively and 6 Months Postoperatively, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No